CLINICAL TRIAL: NCT02491632
Title: Effects of Physical Activity Plus Short Course of Dexamethasone for Cancer-Related Fatigue in Advanced Cancer
Brief Title: Physical Activity and Dexamethasone in Reducing Cancer-Related Fatigue in Patients With Advanced Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2014-0436; NCI-2015-01320 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0436 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-07-03; First posted 2015-07-08 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Neoplasm; Fatigue; Metastatic Malignant Neoplasm; Recurrent Malignant Neoplasm; Refractory Malignant Neoplasm
MeSH Terms: conditions — Fatigue; Neoplasm Metastasis; Recurrence; Neoplasms | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (high-dose dexamethasone, physical activity) (Experimental): Patients receive high-dose dexamethasone PO BID for 7 days. Patients also follow a graded resistance exercise program 3 days a week and a walking regimen at least 5 days a week for 4 weeks. The frequency, duration, and intensity of the exercises will be evaluated and adjusted as necessary.
  Interventions: Drug: Dexamethasone; Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (low dose dexamethasone, physical activity) (Experimental): Patients receive low-dose dexamethasone PO BID for 7 days. Patients also follow a graded resistance exercise program 3 days a week and a walking regimen at least 5 days a week for 4 weeks. The frequency, duration, and intensity of the exercises will be evaluated and adjusted as necessary.
  Interventions: Drug: Dexamethasone; Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Behavioral: Exercise Intervention — Complete a graded resistance exercise program and a walking regimen
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well physical activity and dexamethasone work in reducing cancer-related fatigue in patients with cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced). Dexamethasone is approved for the treatment of tiredness, pain, and nausea. Physical activity may help improve cancer-related fatigue by improvement in symptoms, distress, and overall well-being. It is not yet known whether high dose or low dose dexamethasone combined with physical activity works better in reducing fatigue in patients with advanced cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To determine the feasibility, adherence, and satisfaction with physical activity (PA) plus dexamethasone (PA+ DEX).

SECONDARY OBJECTIVES:

I. To explore the preliminary efficacy of PA+ Hi Dex group (PA for 4 weeks plus high dose dexamethasone for 1 week) and PA + Lo Dex groups (PA for 4 weeks plus low dose dexamethasone for 1 week) on cancer-related fatigue (CRF) as measured by Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) at the end of one week.

II. To explore the effects of PA+ Hi Dex on the various dimensions of CRF (Patient-Reported Outcomes Measurement Information System-Fatigue [PROMIS-F]), i.e., affective/emotional (Hospital Anxiety Depression Scale [HADS]); physical/behavioral (the Multidimensional Fatigue Symptom Inventory-Short Form [MFSI-SF], Pittsburg Sleep Quality Index), physical activity and function (30 second sit-to stand test, six minute walk test) before and after treatment.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive high-dose dexamethasone orally (PO) twice daily (BID) for 7 days. Patients also follow a graded resistance exercise program 3 days a week and a walking regimen at least 5 days a week for 4 weeks. The frequency, duration, and intensity of the exercises will be evaluated and adjusted as necessary.

ARM II: Patients receive low-dose dexamethasone PO BID for 7 days. Patients also follow a graded resistance exercise program 3 days a week and a walking regimen at least 5 days a week for 4 weeks. The frequency, duration, and intensity of the exercises will be evaluated and adjusted as necessary.

After completion of study, patients are followed up at day 29 and again after 1 month.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of advanced cancer (defined as metastatic or recurrent) with fatigue >= 4/10 (0-10 scale) on the Edmonton Symptom Assessment Scale (ESAS)
* The presence of fatigue for at least 2 weeks
* Normal cognition
* Hemoglobin > 8 g/L within 1 week of enrollment in the study
* A life expectancy of >= 4 months
* No evidence of significant anxiety or depression as determined by a total HADS scores of < 21
* Definition of advanced cancer includes those patients who have metastatic or refractory disease according to their treating oncologist
* Patients must be able to understand, read, write, and speak English or Spanish

Exclusion Criteria:

* Patients with a history of hypersensitivity to dexamethasone or having any contraindication to physical activity as determined by the treating physician
* Reports a fall in the past 30 days
* Uncontrolled diabetes mellitus as defined by a random blood sugar of > 200 mg/dl not being monitored by their primary care physician
* Sepsis and/or acute, chronic, or ongoing infections that are currently being treated with systemic antimicrobials
* Will exclude patients with current, active peptic ulcer disease
* Neutropenia as defined by an absolute neutrophil count (ANC) of < 1000 cells/mm
* Regular participation in moderate- or vigorous-intensity physical activity for >= 30 minutes at least 5 times a week and strength training for >= 2 days
* Severe cardiac disease (New York Heart Association functional class III or IV) or coronary artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yennurajalingam S, Valero V, Lu Z, Liu DD, Busaidy NL, Reuben JM, Diaz Fleming C, Williams JL, Hess KR, Basen-Engquist K, Bruera E. Combination Therapy of Physical Activity and Dexamethasone for Cancer-Related Fatigue: A Phase II Randomized Double-Blind Controlled Trial. J Natl Compr Canc Netw. 2021 Dec 29;20(3):235-243. doi: 10.6004/jnccn.2021.7066. PMID 34965510
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from MD Anderson Cancer Center outpatients clinic for supportive are who has a diagnosis of advanced cancer with average intensity of fatigue of >=4/10 on the ESAS scale in the previous 24 hours and presence of fatigue for at least 2 weeks.
Pre-assignment Details: A total of 90 patients were enrolled for this study. Of them 7 withdrew their consent, Doctor did not allow Dexamethasone for 3 cases, 2 had disease progression, and for 2 cases, their oncologist did not approve it. Thus a total of 76 participants were randomized.
Groups:
- Physical Exercise + Low Dose Dexamethasone: Received stabdardizex Physical activity for 4 weeks and 4mg of Dexamethasone orally twice daily for 7 days
- Physical Exercise + High Dose Dexamethasone: Received stabdardizex Physical activity for 4 weeks and 8mg of Dexamethasone orally twice daily for 7 days
Period: Overall Study
Arm/Group | Physical Exercise + Low Dose Dexamethasone | Physical Exercise + High Dose Dexamethasone
Started | 38 | 38
Completed | 31 | 29
Not Completed | 7 | 9

BASELINE CHARACTERISTICS:
Population: Participants who completed the intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Exercise + Low Dose Dexamethasone | Physical Exercise + High Dose Dexamethasone | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [55 to 68] | 58 [53 to 63] | 60 [54 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 28 | 26 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 28 | 27 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60
Cancer Diagnosis [Count of Participants; unit: Participants]
  Breast | 7 | 7 | 14
  Lung | 4 | 3 | 7
  Gastrointestinal | 9 | 5 | 14
  Genitourinary | 8 | 6 | 14
  Other | 3 | 8 | 11
Assessment [Median (Inter-Quartile Range); unit: units on a scale] — Edmonton Symptom Assessment System (ESAS) Fatigue score ranges from 0-10, higher score indicates higher fatigue. Hospital Anxiety and Depression Scale (HADS) Anxiety scores ranges from 0-21, higher score indicates higher anxiety. Hospital Anxiety and Depression Scale (HADS) Depression score ranges from 0-21, higher score indicates higher depression. Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) subscale score ranges from 0-52, lower score indicates higher fatigue.
  units on a scale
    Edmonton Symptom Assessment System (ESAS) Fatigue Score | 6 [5 to 8] | 6 [5 to 7] | 6 [5 to 7.5]
    Hospital Anxiety and Depression Scale (HADS) Anxiety | 4 [2 to 8] | 5 [4 to 8] | 5 [3 to 8]
    Hospital Anxiety and Depression Scale (HADS) Depression | 6 [3 to 8] | 7 [5 to 8] | 6 [4 to 8]
    Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) subscale | 23 [18 to 29.3] | 20 [15 to 31] | 21 [16 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Levels at Day 8 and Day 29
Description: FACIT-F (Functional Assessment of Chronic Illness Therapy-Fatigue) subscale is a 13 item subscale of FACT-G that allows patient to rate the intensity of their fatigue and its related symptoms on a scale of 0 (not at all) to 4 (very much). The total calculated score varied from 0-52 with a lower score indicating a more severe fatigue level. We measured the change in FACIT-F levels between Baseline and Day 8, and between Baseline and Day 29 using Wilcoxon signed rank test.
Time Frame: Baseline, day 8, day 29
Population: Participants who completed the intervention.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Physical Exercise + Low Dose Dexamethasone | Physical Exercise + High Dose Dexamethasone
Number analyzed (Participants) | 31 | 29
score on a scale
  Change between Baseline and Day 8 | 9 [3 to 19] | 8 [3 to 18]
  Change between Baseline and Day 29 | 10 [4 to 16] | 12 [7 to 20]
Statistical Analysis 1: Comparison: Physical Exercise + Low Dose Dexamethasone; Change between Baseline and Day 8; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Physical Exercise + Low Dose Dexamethasone; Change between Baseline and Day 29; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Physical Exercise + High Dose Dexamethasone; Change between Baseline and Day 8; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Physical Exercise + High Dose Dexamethasone; Change between Baseline and Day 29; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System-Fatigue (PROMIS-F) Total
Description: The PROMIS-F (Patient Reported Outcome Measurement Information System-Fatigue) short form was used to measure the experience of fatigue in patients' daily activities over the past week. It consists of 7 items with response options on a 5-point Likert scale, ranging from 1 (never) to 5 (always). We measured the change in PROMIS-F score between Baseline and Day 8, and between Baseline and Day 29 using Wilcoxon signed rank test. The total score is used in the analysis and is obtained by summing keyed scores of all items. Scores can range from 7 to 35, with higher scores indicating greater fatigue.
Time Frame: Baseline, day 8, day 29
Population: Participants who completed the intervention.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Physical Exercise + Low Dose Dexamethasone | Physical Exercise + High Dose Dexamethasone
Number analyzed (Participants) | 31 | 29
units on a scale
  Change between Baseline and Day 8 | -3 [-8 to 0] | -4 [-8 to 0]
  Change between Baseline and Day 29 | -9 [-20 to 0] | -7 [-9 to -1]
Statistical Analysis 1: Comparison: Physical Exercise + Low Dose Dexamethasone; Change between Baseline and Day 8; Test type: Other; p = .003, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Physical Exercise + Low Dose Dexamethasone; Change between Baseline and Day 29; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Physical Exercise + High Dose Dexamethasone; Change between Baseline and Day 8; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Physical Exercise + High Dose Dexamethasone; Change between Baseline and Day 29; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Edmonton Symptom Assessment Scale (ESAS) Fatigue
Description: ESAS (Edmonton Symptom Assessment Scale) is a validated scale ranging from 0 (not at all) to 10 (very much) used to assess 10 symptoms commonly experienced by cancer patients during the previous 24 hours: pain, fatigue, nausea, depression, anxiety, drowsiness, dyspnea, anorexia, sleep and feeling of wellbeing. We measured the change in ESAS fatigue score between Baseline and Day 8, and between Baseline and Day 29 using Wilcoxon signed rank test. Total ESAS fatigue score ranges from 0-10, with a higher score indicating higher fatigue.
Time Frame: Baseline, day 8, day 29
Population: Participants who completed the intervention.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Physical Exercise + Low Dose Dexamethasone | Physical Exercise + High Dose Dexamethasone
Number analyzed (Participants) | 31 | 29
score on a scale
  Change between Baseline and Day 8 | -1.5 [-3 to 0] | -2 [-3 to 0]
  Change between Baseline and Day 29 | -1.5 [-5 to 0] | -3 [-4 to -1]
Statistical Analysis 1: Comparison: Physical Exercise + Low Dose Dexamethasone; Change between Baseline and Day 8; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Physical Exercise + Low Dose Dexamethasone; Change between Baseline and Day 29; Test type: Other; p < .065, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Physical Exercise + High Dose Dexamethasone; Change between Baseline and Day 8; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Physical Exercise + High Dose Dexamethasone; Change between Baseline and Day 29; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Multidimensional Fatigue Symptom Inventory-Short Form (MFSI_SF) Total Score
Description: The MFSI-SF is a 30-item scale used to assess the multidimensional nature of fatigue. Responses are selected using a 5-point scale, ranging from 0 (not at all) to 4 (extremely fatigue). It consists of 5 subscales: general fatigue, physical fatigue, emotional fatigue, mental fatigue and vigor. The MFSI-SF total score is the sum of the general fatigue, physical fatigue, emotional fatigue and mental fatigue subscale score and subtracting vigor subscale score. Thus MFSI-SF total score ranges from 24-96, with a higher score indicating a higher fatigue level. We measured the change in MFSI-SF total score between Baseline and Day 8, and between Baseline and Day 29 using Wilcoxon signed rank test.
Time Frame: Baseline, day 8, day 29
Population: Participants who completed the intervention.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Physical Exercise + Low Dose Dexamethasone | Physical Exercise + High Dose Dexamethasone
Number analyzed (Participants) | 31 | 29
score on a scale
  Change between Baseline and Day 8 | -9 [-16 to -3] | -5 [-16 to 3]
  Change between Baseline and Day 29 | -6 [-10 to -1] | -4.5 [-15.5 to 6.5]
Statistical Analysis 1: Comparison: Physical Exercise + Low Dose Dexamethasone; Change between Baseline and Day 8; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Physical Exercise + Low Dose Dexamethasone; Change between Baseline and Day 29; Test type: Other; p = .30, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Physical Exercise + High Dose Dexamethasone; Change between Baseline and Day 8; Test type: Other; p = .19, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Physical Exercise + High Dose Dexamethasone; Change between Baseline and Day 29; Test type: Other; p = .27, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 29
Arm/Group | Physical Exercise + Low Dose Dexamethasone | Physical Exercise + High Dose Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/31 | 1/29
Serious Adverse Events (participants affected / at risk) | 5/31 | 4/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Physical Exercise + Low Dose Dexamethasone (N=31) | Physical Exercise + High Dose Dexamethasone (N=29)
Eye Infection (Eye disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Kidney Infection (Infections and infestations) | 1 | 1
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Thromboembolic Event (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT02491632/Prot_SAP_000.pdf